CLINICAL TRIAL: NCT01050127
Title: A Study of Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Doses of ABT-436 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Katherine Tracy, MD, PhD, Abbott
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M11-731
Record Dates: First submitted 2009-12-04; First posted 2010-01-15 (Estimated); Last update posted 2010-11-03 (Estimated); Status verified 2010-09

CONDITIONS: Healthy
Keywords: Pharmacokinetics; Pharmacodynamics; Drug Safety; Phase 1 Clinical Trial

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Low dose ABT-436 (Experimental): ABT-436 or placebo administered once daily for 7 days.
  Interventions: Drug: ABT-436; Drug: Placebo
- Mid Dose ABT-436 (Experimental): ABT-436 or placebo administered once daily for 7 days.
  Interventions: Drug: ABT-436; Drug: Placebo
- High Dose ABT-436 (Experimental): ABT-436 or placebo administered once daily for 14 days.
  Interventions: Drug: ABT-436; Drug: Placebo

INTERVENTIONS:
Drug: ABT-436 — See Arm Description for details.
Drug: Placebo — See Arm Description for details.

SUMMARY:
The objectives of this study are to assess the safety, tolerability, pharmacodynamics and pharmacokinetics of multiple doses of ABT-436 in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

1. Age is between 18 and 55 years, inclusive.
2. If female, subject must be postmenopausal for at least two years or surgically sterile.
3. Females must have negative results for pregnancy tests prior to study drug administration.
4. If male, subject must be surgically sterile or agree to be sexually inactive or agree to use a barrier method of birth control.
5. Body Mass Index is 18.0 to 29.9 kg/m2 (2 = superscript number), inclusive.
6. A condition of general good health based upon the results of a medical history, physical examination, vital signs, laboratory profile, and a 12-lead electrocardiogram.
7. Must voluntarily sign and date an informed consent, approved by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB), prior to the initiation of any screening or study-specific procedures.

Exclusion Criteria:

1. History of significant sensitivity or allergy to any drug.
2. Use of known inhibitors or inducers of CYP3A within 30 days prior to the first dose of study drug and through the end of the study.
3. Requirement for, or use of within the 2-week period prior to study drug administration, any over-the-counter or prescription medication, vitamins, minerals or herbal supplements on a regular basis.
4. Receipt of any depot drug by injection within 30 days prior to study drug administration.
5. Positive screen for drugs of abuse or alcohol, or recent (6-month) history of drug or alcohol abuse.
6. Use of tobacco or other nicotine-containing products within the six-month period preceding study drug administration.
7. Donation or loss of 550 mL of blood or more (including plasmapheresis) or receipt of a transfusion of any blood product within 8 weeks prior to the first dose of study drug.
8. Receipt of an investigational product within a time period equal to 10 half-lives, if known, or a minimum of 6 weeks prior to study drug administration.
9. Has a clinically significant abnormal diastolic blood pressure (< 45 or > 90 mm Hg), systolic blood pressure (< 85 or > 140 mm Hg) or heart rate (< 45 or > 100 bpm).
10. HbA1c > 6.0%.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2009-12; Primary Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability Assessments (i.e., electrocardiogram(ECG), clinical laboratory tests, vital signs, weight, adverse events (AE) assessment, pulmonary function tests, physical and brief neurological examinations) | Days -2 through Day 7 or 14
Assess Pharmacokinetics (i.e., ABT-436 and possible metabolite levels) | Day -1 through Day 7
Pharmacodynamics (i.e., biomarkers of drug effect) | Day -1 through Day 7

CONTACTS AND LOCATIONS:
Locations (1):
- Site Reference ID/Investigator# 24849, Waukegan, Illinois, United States